CLINICAL TRIAL: NCT00384553
Title: Risk Adapted Therapy Optimization for Patients With Relapsed or Refractory Aggressive Non-Hodgkin-Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Magdeburg (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSHO #071
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab
Drug: DHAP
Drug: TEC
Drug: autologous stem cell transplantation

SUMMARY:
This study investigates toxicity and efficacy of 2 x R-DHAP followed by High dose chemotherapy R-TEC and autologous stem cell transplantation in patients with relapsed or refractory aggressive Non- Hodgkins's Lymphoma.

DETAILED DESCRIPTION:
Initial Cytoreduction is performed with DHAP- protocol using dexamethasone, cytarabine and cisplatin followed by high dose chemotherapy with treosulfan, etoposide and cisplatin (TEC) an autologous peripheral blood stem cell transplantation(aPBSCT). In case of only partial remission a second identical high dose chemotherapy and aPBSCT follows. Patients with primary refractory disease or early relapse within 6 months should receive a allogenous stem cell transplantation. For Patients with CD 20 positive B-cell lymphoma the chemotherapy regiments DHAP and TEC are combined with rituximab.

ELIGIBILITY:
Inclusion Criteria:

* first relapse or primary refractory disease of aggressive Non-Hodgkin's lymphoma stage I-IV
* pretreatment with systemic therapy
* 18-65 years of age
* Performance status:ECOG 0-2
* Granulocyte count >1.5/µm3, Platelet count >100/µm3
* Creatinine -Clearance ≥ 1 ml/sec
* GPT/GOT ≤ 1.5 x normal (except tumour related)
* Bilirubine < 22 µmol/l
* no participation in another study 3 month before and during this study
* informed consent

Exclusion Criteria:

* Second neoplasia in history or existing except basalioma or squamous epithelium carcinoma of the skin or removed cervical intraepithelial neoplasia
* CNS- involvement by lymphoma
* respiratory Partial- or global insufficiency
* cardiac insufficiency (NYHA-Stage 3-4, EF < 30 %)
* severe neurological or psychiatric disease
* pregnancy
* HIV positivity ,active virus hepatitis, bacterial infection
* No follow up procedures ensured

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-06; Study Completion 2010-06

PRIMARY OUTCOMES:
Toxicity

SECONDARY OUTCOMES:
remission rate
remission duration
overall survival
relapse free survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koenigsmann, PD Dr. med., Principal Investigator — University of Magdeburg
Locations (1):
- University of Magdeburg, Magdeburg, Germany